CLINICAL TRIAL: NCT03777371
Title: Anti-HIV False Positivity Rate in Pregnant Women; and Investigating the Factors Affecting This Situation
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: HIVinPregnancies
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: HIV Seropositivity; Acquired Immunodeficiency Syndrome; Pregnancy, High Risk
MeSH Terms: conditions — HIV Seropositivity; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anti HIV Seropositive Pregnant Women

SUMMARY:
HIV virus is an etiologic agent of ( AIDS ) immunodeficiency syndrome . It is known that the estimated rate of transfer from mother to baby is 25% to 45%, pregnancy rate is 5-10%, pregnancy rate is 15-20% and in lactation period is 5-10%. Risk factors; maternal viral load, breastfeeding, vaginal birth, and prematurity. Although there is a high rate of false positivity in prenatal screening in our country, one of the factors affecting this is the number of pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Anti HIV seropositive Pregnant Women

Exclusion Criteria:

* Anti HIV seronegative Pregnant Women

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women between 8 and 40 weeks of gestation
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The effect of the number of pregnancies on Anti HIV false positivity rate | 5 years

IPD SHARING:
Plan to Share IPD: Yes